CLINICAL TRIAL: NCT05485935
Title: A Confirmatory, Multi-centre, Randomized, Open Label, Controlled Study Confirming Performance of a Single-use Intermittent Micro-holes Zone Catheter in a Population of Adult Male Intermittent Catheter Users.
Brief Title: A Confirmatory Study Confirming Performance of a New Intermittent Catheter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CP334
Record Dates: First submitted 2022-06-30; First posted 2022-08-03 (Actual); Results first posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-02

CONDITIONS: Urinary Retention
MeSH Terms: conditions — Urinary Retention

STUDY DESIGN:
Intervention Model Description: This was a multi-centre, randomized, controlled crossover design. The total study duration for the individual participant was approximately 9 weeks. The study consisted of four study visits (V0-V3) and two 4-week test periods at home (T1 and T2). Visit 0 and 1 was performed on the same day if subjects allowed.
  One population included all enrolled subjects who took part in the two test periods in a home setting only (T1 and T2). This constituted the Full Analysis Set (FAS) 1 (N=73) where only endpoints related to dipstick hematuria, catheter perception and quality of life were assessed.
  A subset of subjects from the FAS1 also took part in two clinic visits (V2 and V3) where endpoints related to bladder emptying and discomfort were assessed. One visit took place in between the two test periods at home (V2) and the other visit took place after the last test period at home (V3) which was also the termination visit. This subset is termed the FAS 2 (N=49).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigational device - intermittent catheter with micro-hole zone (Experimental): Single-use, sterile, hydrophilic coated intermittent male catheter. The external diameter is measured in millimeters (Charrière scale: Ch, CH) and the sizes available were CH12 and CH14 with a flexible tip and a micro-hole zone for urinary drainage.
  Interventions: Device: Investigational device - intermittent catheter with micro-hole zone
- Comparator device - standard intermittent catheter (Active Comparator): Single-use, sterile, hydrophilic coated intermittent male catheters (sizes CH12 and CH14) with sleeves: SpeediCath Flex, VaPro, VaPro Pocket, VaPro Plus and VaPro Plus Pocket.
  Interventions: Device: Comparator - standard intermittent catheter

INTERVENTIONS:
Device: Investigational device - intermittent catheter with micro-hole zone — Intermittent male catheter with micro-hole zone for urinary drainage
  Arms: Investigational device - intermittent catheter with micro-hole zone
Device: Comparator - standard intermittent catheter — SpeediCath Flex, VaPro Pocket, VaPro Plus and VaPro Plus Pocket.
  Arms: Comparator device - standard intermittent catheter

SUMMARY:
A multi-centre, randomized, controlled crossover design. The total study duration for the individual subject was approximately 9 weeks. The study consisted of four study visits (V0-V3) and two 4-week test periods at home (T1 and T2). Visit 0 and 1 was performed on the same day if subjects allowed.

One population included all enrolled subjects who took part in the two test periods in a home setting only (T1 and T2). This constituted the Full Analysis Set (FAS) 1 (N=73)where only endpoints related to dipstick hematuria, catheter perception and quality of life were assessed.

A subset of subjects from the FAS1 also took part in two clinic visits (V2 and V3) where endpoints related to bladder emptying and discomfort were assessed. One visit took place in between the two test periods at home (V2) and the other visit took place after the last test period at home (V3) which was also the termination visit. This subset is termed the FAS 2 (N=49).

DETAILED DESCRIPTION:
This investigation was a multi-centre, randomized, controlled crossover study including 73 male clean intermittent catheterization (CIC) users.

The study consisted of four study visits (V0-V3) and two 4-week test periods at home (T1 and T2). Visit 0 and 1 were performed on the same day if participants allowed. Visit 0 included the screening-, inclusion-, and randomization phase of participants and at visit 1, participants performed a self-catheterization with the device according to their respective randomization scheme. This was followed by a dipstick test for hematuria. This constituted the Full Analysis Set (FAS) 1, consisting of 73 participants.

In the two 4-week test periods (T1 and T2, respectively) the participants catheterized at home with the specified catheter according to their randomization scheme. Both 4-week periods started with a 2-week run-in period followed by a 2-week period during which a dipstick test for hematuria was performed daily.

For Visit 2 and 3, a sub-group of participants was invited for a clinical test visit during which participants were catheterized with the same device applied during the preceding home-test period. First a healthcare professional (HCP)-led catheterization was performed followed by a self-catheterization, and endpoints related to bladder emptying (residual urine and number of urinary flow-stop episodes) were measured. After each catheterization, any residual urine left in the bladder was measured with a bladder scanner and hematuria was assessed with a dip-stick test. After the self-catheterization process, subjects at clinic visit V2 and V3 completed a questionnaire related to discomfort.This constituted the Full Analysis Set (FAS) 2, consisting of 49 participants.

All participants completed a perception questionnaire and a HRQoL questionnaire associated with the catheter during the last two weeks of the home test period. For participants not part of clinic visits V2 and V3, a nurse assisted with the questionnaires after each home-test period during a remote home visit. Thereafter, all participants were introduced to the second device to be tested for the next home-test period.

After the second home-test period, the study was terminated with a test visit 3 (V3), either in the clinic (for the subset group, FAS2) or a home visit by the nurse (the FAS1 group).

ELIGIBILITY:
Inclusion Criteria:

1. Male
2. Was at least 18 years of age and had full legal capacity
3. Had given written informed consent
4. Had signed letter of authority (only DK)
5. Had used clean intermittent self-catheterization (CISC) for at least the last 3 months
6. Had used intermittent catheterization as the only bladder emptying method for at least the last 3 months
7. Self-catheterized using Coloplast SpeediCath Flex or Hollister VaPro catheters, CH12 or CH14, for at least 3 months prior to inclusion
8. Had the ability (assessed by investigator) and willingness to adhere to a 2-month study period

Exclusion Criteria

1. Participation in any other clinical study during this investigation
2. Previous participation in the study
3. Symptoms of urinary tract infection as judged by the investigator (rescheduling allowed within recruitment period for LPI)
4. Individuals with history, suspected or showing signs of producing urine with excessive amount of mucus or large/clustered sediments or debris
5. Any known allergies towards ingredients in the investigational device

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male users of intermittent urinary catheterizations to empty their bladder.
Enrollment: 73 (Actual)
Dates: Start 2022-08-20 (Actual); Primary Completion 2023-01-03 (Actual); Study Completion 2023-01-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nikesh thiruchelvam, Dr, Study Chair — NHS Foundation Trust
Locations (6):
- Denmark (2):
  - Sanos Clinic, Gandrup, North Denmark
  - Rigshospitalet, Copenhagen
- France (2):
  - Hopital Claude Huriez, Lille
  - Hôpital Tenon, Paris
- Artimed, Kassel, Germany
- Illingworth Research Group, Macclesfield, Cheshire, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Investigational Device (Intermittent Catheter With Micro-hole Zone, CH12 or CH14) Then Comparator: Participants were randomly assigned to the sequence of two intervention arms, in block sizes of 8.
  During the first period, participants were catheterized with the investigational device during a first clinic visit, followed by a 4 weeks period of home catheterization. A sub-population were invited for a second clinic visit (V2) and were catheterized with the investigational device by an HCP and a self-catheterization, respectively.
  At the second intervention period, participants catheterized with the comparator device during another 4 weeks at home. The same sub-population took part in a third and final clinic visit (V3) and were catheterized by a HCP- and a self-catheterization, respectively.
- Comparator Device (Standard Intermittent Catheter, CH12/14) Then Investigational Device: Participants were randomly assigned to the sequence of two intervention arms, in block sizes of 8.
  During the first period, participants were catheterized with the comparator device during a first clinic visit (V1), followed by a 4 weeks period of home catheterization. A sub-population were invited for a second clinic visit (V2) and were catheterized with the comparator device by an HCP and a self-catheterization, respectively.
  At the second intervention period, participants catheterized with the investigational device during another 4 weeks at home. The same sub-population took part in a third and final clinic visit (V3) and were catheterized by a HCP- and a self-catheterization, respectively.
Period: Period 1 (V0, V1, T1, and V2)
Arm/Group | Investigational Device (Intermittent Catheter With Micro-hole Zone, CH12 or CH14) Then Comparator | Comparator Device (Standard Intermittent Catheter, CH12/14) Then Investigational Device
Started | 36 | 37
Completed | 32 | 36
Not Completed | 4 | 1
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 3 | 0
Period: Period 1 (V2 Subpopulation)
Arm/Group | Investigational Device (Intermittent Catheter With Micro-hole Zone, CH12 or CH14) Then Comparator | Comparator Device (Standard Intermittent Catheter, CH12/14) Then Investigational Device
Started | 23 (A subpopulation of at least 42 participants were invited for clinic visits to test the catheter performance) | 26 (A subpopulation of at least 42 participants were invited for clinic visits to test the catheter performance)
Completed | 23 | 26
Not Completed | 0 | 0
Period: Period 2 (T2 and V3)
Arm/Group | Investigational Device (Intermittent Catheter With Micro-hole Zone, CH12 or CH14) Then Comparator | Comparator Device (Standard Intermittent Catheter, CH12/14) Then Investigational Device
Started | 32 | 36
Completed | 32 | 34
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 1
Not completed — loss of contact | 0 | 1
Period: Period 2 (V3 Subpopulation)
Arm/Group | Investigational Device (Intermittent Catheter With Micro-hole Zone, CH12 or CH14) Then Comparator | Comparator Device (Standard Intermittent Catheter, CH12/14) Then Investigational Device
Started | 23 | 26
Completed | 23 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total ITT Population Baseline Measures: As this study was a crossover study, each participant underwent catheterizations with both the investigational device and the comparator device. The study consisted of four study visits (V0-V3) and two 4-week test periods at home (T1 and T2). Visit 0 included subject screening, enrollment, and randomization. Randomization was done centralized, randomly assigning subjects to two intervention sequences in block-sizes of four. Hence, the first group was catheterized with the investigational device at visit 0 and 1, followed by a test period at home (T1) and a follow-up visit (V2). Subsequently, the comparator device was tested during the next test period at home (T2) followed by a visit 3 which also terminated the study. The second group tested the devices in reversed order. The total study duration was approximately nine weeks for the individual subject
Arm/Group | Total ITT Population Baseline Measures
Number analyzed (Participants) | 73
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.9 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 73
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Denmark | 46
  United Kingdom | 13
  France | 6
  Germany | 8
Number of participants with neurogenic bladder dysfunction [Count of Participants; unit: Participants] | 28
Number of participants with non-neurogenic bladder dysfunction [Count of Participants; unit: Participants] | 45

OUTCOME MEASURES:

1. Primary Outcome: Residual Urine at 1st Flow Stop (HCP-led Catheterization) i.e., Total Catheterisation Volume Minus Volume at 1st Flow-stop, Both Derived From a Catheterisation Profile
Description: The residual urine at 1st flow-stop during catheterization (performed by a HCP) represents the volume of urine left in the bladder, the first time the urine stops running out of the catheter during bladder emptying.
  Hence, the residual volume at 1st flow-stop was calculated as the total volume post catheterisation minus the volume at 1st flow-stop, derived from a catheterisation profile which was connected to a time-logged weighing [g].
Time Frame: Immediately after the procedure/catheterization, at second and third clinic visit following 4 weeks of home catheterization
Population: This population constituted a subset (=Full Analysis Set 2(FAS2)) of the all randomized subjects (FAS1, N=73). This subset FAS2 included 49 participant, who took part in both test periods at home (T1 and T2) and in clinic visits (V2 and V3) to acquire data related to the catheterization process and which supported the primary endpoints residual urine at first flow-stop and number of flow-stop episodes.
Measure: Mean (95% Confidence Interval); unit: mL
Groups:
- Investigational Device (Intermittent Catheter With Micro-hole Zone, CH12 or CH14): Participants were randomly assigned to the sequence of two intervention arms, in block sizes of 8.
  At the first intervention, one catheterization was performed with the investigational during a first clinic visit, followed by a 4 weeks period of home catheterization, followed by a second clinic visit with a HCP- and a self-catheterization, respectively.
  At the second intervention, catheterizations with the comparator device were performed during a second 4 weeks period at home, followed by a third and final clinic visit with a HCP- and a self-catheterization, respectively.
- Comparator Device (Standard Intermittent Catheter, CH12/14): Participants were randomly assigned to the sequence of two intervention arms, in block sizes of 8.
  At the first intervention, one catheterization was performed with the comparator during a first clinic visit, followed by a 4 weeks period of home catheterization, followed by a second clinic visit with a HCP- and a self-catheterization, respectively.
  At the second intervention, catheterizations with the investigational device were performed during a second 4 weeks period at home, followed by a third and final clinic visit with a HCP- and a self-catheterization, respectively.
Arm/Group | Investigational Device (Intermittent Catheter With Micro-hole Zone, CH12 or CH14) | Comparator Device (Standard Intermittent Catheter, CH12/14)
Number analyzed (Participants) | 49 | 49
mL | 18 [7.05 to 28.94] | 63.93 [37.86 to 90.01]
Statistical Analysis 1: Comparison: Investigational Device (Intermittent Catheter With Micro-hole Zone, CH12 or CH14) vs Comparator Device (Standard Intermittent Catheter, CH12/14); This was a superiority investigation in which the null hypothesis of the primary endpoints was to be rejected, at a 5% significance (alpha 0.05), to demonstrate the superiority of the investigational device; Test type: Superiority; p = 0.001, Mixed Models Analysis — The pass criteria were based on results analysing the 2 primary endpoints in a hierarchical fashion: rejecting the H0 on the first endpoint (Residual urine at first flow-stop) before continuing to the second (Number of flow-stop episodes); Mean Difference (Final Values) = 45.94, 95% CI 2-sided [19.24 to 72.64]

2. Primary Outcome: Number of Flow-stop Episodes (HCP-led Catheterization)
Description: Number of flow-stop episodes were determined as instances where the flow rate decreased to less than 0.8 mL/s for a period of at least two seconds. All episodes were detected by automatic thresholding, followed by manual inspection, where the intra-catheter pressure readings were used to support the assessment of a flow stop.
Time Frame: Immediately after catheterisation, at second and third clinic visit following 4 weeks of home catheterization
Population: This population constituted a subset (= Full analysis set (FAS)2) of the all randomized subjects (FAS1, N=73). This subset FAS2 included 49 participant, who took part in both test periods at home (T1 and T2) and in clinic visits (V2 and V3) to acquire data related to the catheterization process and which supported the primary endpoints residual urine at first flow-stop and number of flow-stop episodes.
Measure: Mean (95% Confidence Interval); unit: Flow stop episodes
Arm/Group | Investigational Device (Intermittent Catheter With Micro-hole Zone, CH12 or CH14) | Comparator Device (Standard Intermittent Catheter, CH12/14)
Number analyzed (Participants) | 49 | 49
Flow stop episodes | 0.20 [0.09 to 0.43] | 1.32 [0.96 to 1.80]
Statistical Analysis 1: Comparison: Investigational Device (Intermittent Catheter With Micro-hole Zone, CH12 or CH14) vs Comparator Device (Standard Intermittent Catheter, CH12/14); [analysis description as in outcome 1, analysis 1]; Test type: Superiority — The pass criteria were based on the results analysing the two primary endpoints in a hierarchical fashion: rejecting the null hypothesis on the first endpoint (Residual urine at first flow-stop) before continuing to the second (Number of flow-stop episodes); p < 0.001, Mixed Models Analysis; Risk Ratio (RR) = 0.15, 95% CI 2-sided [0.07 to 0.35]

3. Secondary Outcome: Number of Flow-stop Episodes (Self-led Catheterization)
Description: Number of flow-stops were measured with a pressure sensor, which is an electronic device used for monitoring the hydrostatic pressure at the outlet of an intermittent urinary catheter during emptying. From a sensor curve, flow-stops were identified by two individually trained evaluators as a hydrostatic pressure peak coinciding with a urine flow-stop/ urine dripping (flowrate lower than 0,8 ml/sec). Results from both evaluators were compared and in case of discrepancy a discussion was performed to extenuate discrepancies and agree on a final interpretation of the curves.
Time Frame: as for outcome 1
Population: This population constituted a subset (FAS2) of the all randomized subjects (FAS1, N=73). This subset FAS2 included 49 participant, who took part in both test periods at home (T1 and T2) and in clinic visits (V2 and V3) to acquire data related to the catheterization process and which supported the primary endpoints residual urine at first flow-stop and number of flow-stop episodes.
Measure: Mean (95% Confidence Interval); unit: Flow stop episodes
Groups:
- Investigational Device (Intermittent Catheter With Micro-hole Zone, CH12 or CH14) Then Comparator: Participants were randomly assigned to the sequence of two intervention arms, in block sizes of 8.
  At the first intervention, one catheterization was performed with the investigational during a first clinic visit, followed by a 4 weeks period of home catheterization, followed by a second clinic visit with a HCP- and a self-catheterization, respectively.
  At the second intervention, catheterizations with the comparator device were performed during a second 4 weeks period at home, followed by a third and final clinic visit with a HCP- and a self-catheterization, respectively.
- Comparator Device (Standard Intermittent Catheter, CH12/14) Then Investigational Device: Participants were randomly assigned to the sequence of two intervention arms, in block sizes of 8.
  At the first intervention, one catheterization was performed with the comparator during a first clinic visit, followed by a 4 weeks period of home catheterization, followed by a second clinic visit with a HCP- and a self-catheterization, respectively.
  At the second intervention, catheterizations with the investigational device were performed during a second 4 weeks period at home, followed by a third and final clinic visit with a HCP- and a self-catheterization, respectively.
Arm/Group | Investigational Device (Intermittent Catheter With Micro-hole Zone, CH12 or CH14) Then Comparator | Comparator Device (Standard Intermittent Catheter, CH12/14) Then Investigational Device
Number analyzed (Participants) | 49 | 49
Flow stop episodes | 0.13 [0.04 to 0.37] | 0.96 [0.65 to 1.43]
Statistical Analysis 1: Comparison: Investigational Device (Intermittent Catheter With Micro-hole Zone, CH12 or CH14) Then Comparator vs Comparator Device (Standard Intermittent Catheter, CH12/14) Then Investigational Device; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p < 0.001, Mixed Models Analysis; Risk Ratio (RR) = 0.13, 95% CI 2-sided [0.04 to 0.40]

4. Secondary Outcome: Residual Urine at 1st Flow Stop (Self-led Catheterization)
Description: The residual urine at 1st flow-stop during catheterization (performed by the participant self) represents the volume of urine left in the bladder, the first time the urine stops running out of the catheter during bladder emptying.
  Hence, the residual volume at 1st flow-stop was calculated as the total volume post catheterisation minus the volume at 1st flow-stop, derived from a catheterisation profile which was connected to a time-logged weighing [g].
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: mL
Arm/Group | Investigational Device (Intermittent Catheter With Micro-hole Zone, CH12 or CH14) | Comparator Device (Standard Intermittent Catheter, CH12/14)
Number analyzed (Participants) | 49 | 49
mL | 8.2 [-5.6 to 22.1] | 36.8 [23.1 to 50.05]
Statistical Analysis 1: Comparison: Investigational Device (Intermittent Catheter With Micro-hole Zone, CH12 or CH14) vs Comparator Device (Standard Intermittent Catheter, CH12/14); [analysis description as in outcome 1, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.004, Mixed Models Analysis; Mean Difference (Final Values) = 28.5, 95% CI 2-sided [9.5 to 47.6]

5. Secondary Outcome: Mean Red Blood Cell Concentration
Description: The average (mean) Red blood cell concentration based on a dipstick test, collected daily during the two weeks of the home test period T1 and T2 [Erythrocytes/µL].
Time Frame: Dipstick test for haematuria was performed daily were performed in week 3 and 4 (1st home-period) and in week 7 and 8 (2nd home-period).
Population: Participants from the full analysis set during the first and second home period (FAS1)
Measure: Least Squares Mean (95% Confidence Interval); unit: erythrocytes per microliter
Arm/Group | Investigational Device (Intermittent Catheter With Micro-hole Zone, CH12 or CH14) | Comparator Device (Standard Intermittent Catheter, CH12/14)
Number analyzed (Participants) | 66 | 66
erythrocytes per microliter | 16.25 [6.69 to 25.81] | 19.77 [10.20 to 29.33]

6. Secondary Outcome: Positive Hematuria Event Post-catheterisation
Description: Number of positive hematuria events (i.e., blood in urine) based on a dipstick test, collected daily during the final two weeks of the home test period T1 and T2 [positive/negative scale]. Positive value = blood in the urine. Negative value = no blood in the urine.
Time Frame: week 3 and 4 (1st home-period) and in week 7 and 8 (2nd home-period).
Population: Participants from the full analysis set during the first and second home period, (FAS1).
Measure: Mean (95% Confidence Interval); unit: positive hematuria events
Arm/Group | Investigational Device (Intermittent Catheter With Micro-hole Zone, CH12 or CH14) | Comparator Device (Standard Intermittent Catheter, CH12/14)
Number analyzed (Participants) | 66 | 66
positive hematuria events | 0.17 [0.14 to 0.19] | 0.19 [0.17 to 0.22]

ADVERSE EVENTS:
Time Frame: The study consisted of four study visits in a clinic (V0-V3) and two 4-week test periods at home. Hence, the total study duration for the individual subject lasted approximately nine weeks.
Groups:
- Investigational Device; Comparator Device: As this study was a crossover study, each participant underwent catheterizations with both the investigational device and the comparator device.
  Safety population constitutes the full analysis set.
Arm/Group | Investigational Device | Comparator Device
All-Cause Mortality (participants affected / at risk) | 0/73 | 1/73
Serious Adverse Events (participants affected / at risk) | 3/73 | 0/73
Other Adverse Events (participants affected / at risk) | 8/73 | 8/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Investigational Device (N=73) | Comparator Device (N=73)
Cardiac arrest (Cardiac disorders) | 1 (1) | NA
Urosepsis (Renal and urinary disorders) | 1 (1) | NA
unbalanced type 2 diabetes (Endocrine disorders) | 1 (1) | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Investigational Device (N=73) | Comparator Device (N=73)
Urinary tract infection (Renal and urinary disorders) | 2 (2) | 2 (2)
Fever (Infections and infestations) | 1 (1) | 0 (0)
Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Urolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Epididymit (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Blood in urine (Renal and urinary disorders) | 1 (1) | 0 (0)
Gout (Infections and infestations) | 0 (0) | 1 (1)
Swollen foot (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Stinging in urethra (Renal and urinary disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Micturition (Renal and urinary disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-21): https://cdn.clinicaltrials.gov/large-docs/35/NCT05485935/Prot_SAP_000.pdf